CLINICAL TRIAL: NCT03240588
Title: NAVITAS and ENVISION Study: A Study to Characterize the Relationship Between Select Objective Metrics and Clinical Outcomes in Chronic Pain Patients Treated With Boston Scientific Neurostimulation Systems
Brief Title: NAVITAS and ENVISION - Study to Characterize Select Objective Metrics & Clinical Outcomes in Chronic Pain Patients With Boston Scientific Neurostimulation Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 92100126; 92366204 (Other: Boston Scientific protocol number)
Record Dates: First submitted 2017-07-11; First posted 2017-08-07 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study (Experimental): Patients enrolled in the ENVISION study. Follow-up period is based on date they signed the informed consent and were enrolled into the study.
  All commercially approved Boston Scientific neurostimulation systems indicated for the treatment of chronic pain, except for Precision™ and Precision™ Plus.
  Interventions: Device: Neurostimulation System
- Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 SCS Trial Procedure) Navitas Study (Experimental): Patients enrolled in the NAVITAS study. Follow-up period is based on date of their SCS Trial Procedure.
  All commercially approved Boston Scientific neurostimulation systems indicated for the treatment of chronic pain.
  Interventions: Device: Neurostimulation System
- Boston Scientific SCS Systems (Day 0 Implantable Pulse Generator (IPG) Activation) Navitas Study (Experimental): Patients enrolled in the NAVITAS study. Follow-up period is based on date of their Implantable Pulse Generator (IPG) was activated.
  All commercially approved Boston Scientific neurostimulation systems indicated for the treatment of chronic pain.
  Interventions: Device: Neurostimulation System

INTERVENTIONS:
Device: Neurostimulation System — Spinal cord stimulation

SUMMARY:
The objective of the study is to characterize the relationship between select objective metrics and clinical outcomes in chronic pain patients treated with Boston Scientific commercially approved neurostimulation systems.

ELIGIBILITY:
Key Inclusion Criteria:

- Is willing and able to comply with completing protocol required assessments and evaluations

Key Exclusion Criteria:

- Has any pain-related diagnosis, medical/psychological condition or external factors that, in the investigator's medical judgment, might confound reporting of study outcomes (e.g. history of pelvic pain, anginal pain, chronic migraine, involved in litigation, workmen's compensation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, M.S., Study Director — Boston Scientific Neuromodulation Corporation
Locations (16):
- United States (16):
  - Hope Research Institute, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Coastal Research Institute, Carlsbad, California
  - South Lake Pain Institute, Inc, Clermont, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - Tallahassee Neurological Clinic, PA, Tallahassee, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Willis-Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - Forest Health Medical Center, Ypsilanti, Michigan
  - KC Pain Centers, Lee's Summit, Missouri
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Precision Spine Care, Tyler, Texas
  - Washington Center for Pain Management, Bellevue, Washington
  - EvergreenHealth Pain Care, Kirkland, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study: Patients enrolled in the ENVISION study. Follow-up period is based on date they signed the informed consent and were enrolled into the study.
  All commercially approved Boston Scientific neurostimulation systems indicated for the treatment of chronic pain, except for Precision™ and Precision™ Plus.
  Neurostimulation System: Spinal cord stimulation
- Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 SCS Trial Procedure) Navitas Study: Patients enrolled in the NAVITAS study. Follow-up period is based on date of their SCS Trial Procedure.
  All commercially approved Boston Scientific neurostimulation systems indicated for the treatment of chronic pain.
  Neurostimulation System: Spinal cord stimulation
- Boston Scientific SCS Systems (Day 0 Implantable Pulse Generator (IPG) Activation) Navitas Study: Patients enrolled in the NAVITAS study. Follow-up period is based on date of their Implantable Pulse Generator (IPG) was activated.
  All commercially approved Boston Scientific neurostimulation systems indicated for the treatment of chronic pain.
  Neurostimulation System: Spinal cord stimulation
Period: Overall Study
Arm/Group | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 SCS Trial Procedure) Navitas Study | Boston Scientific SCS Systems (Day 0 Implantable Pulse Generator (IPG) Activation) Navitas Study
Started | 363 | 150 | 31
Completed | 178 | 54 | 21
Not Completed | 185 | 96 | 10
Not completed — Death | 3 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 0
Not completed — Lost to Follow-up | 9 | 4 | 0
Not completed — Physician Decision | 3 | 2 | 0
Not completed — Did not meet eligibility criteria | 0 | 6 | 0
Not completed — No longer meets protocol criteria | 12 | 7 | 0
Not completed — Withdrawal by Subject | 60 | 52 | 7
Not completed — Other, additional details not available. | 0 | 12 | 1
Not completed — Attempted to implant study device but unable to do so/unsuccessful neurostimulation trial procedure | 14 | 3 | 0
Not completed — Closure of study | 55 | 3 | 0
Not completed — Subject non-compliance | 23 | 2 | 1
Not completed — Device Deficiency | 1 | 0 | 0
Not completed — End of study information not provided to determine reason for withdrawal. | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Data is based on all available data. More subjects in the "Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study" Arm/Group completed the Baseline outcome measure and Region of Enrollment (359) than the Age and Sex Baseline measures which had 298 patients and the Race/Ethnicity which had 304.
Groups:
- Total: Total of all reporting groups
Arm/Group | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 SCS Trial Procedure) Navitas Study | Boston Scientific SCS Systems (Day 0 Implantable Pulse Generator (IPG) Activation) Navitas Study | Total
Number analyzed (Participants) | 359 | 149 | 31 | 539
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Data is based on all available data. More subjects in the "Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study" Arm/Group completed the Baseline outcome measure and Region of Enrollment (359) than the Age and Sex Baseline measures which had 298 patients and the Race/Ethnicity which had 304.
  years
    Age: number analyzed (Participants) | 298 | 149 | 31 | 478
    Age | 61.2 (11.7) | 58.6 (12.5) | 60.1 (10.4) | 60.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data is based on all available data. More subjects in the "Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study" Arm/Group completed the Baseline outcome measure and Region of Enrollment (359) than the Age and Sex Baseline measures which had 298 patients and the Race/Ethnicity which had 304.
  Participants
    number analyzed (Participants) | 298 | 149 | 31 | 478
    Female | 181 | 97 | 18 | 296
    Male | 117 | 52 | 13 | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data is based on all available data. More subjects in the "Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study" Arm/Group completed the Baseline outcome measure and Region of Enrollment (359) than the Age and Sex Baseline measures which had 298 patients and the Race/Ethnicity which had 304.
  Participants
    American Indian or Alaska native: number analyzed (Participants) | 304 | 149 | 31 | 484
    American Indian or Alaska native | 2 | 2 | 1 | 5
    Asian: number analyzed (Participants) | 304 | 149 | 31 | 484
    Asian | 0 | 0 | 0 | 0
    Black, of African heritage: number analyzed (Participants) | 304 | 149 | 31 | 484
    Black, of African heritage | 19 | 14 | 5 | 38
    Caucasian: number analyzed (Participants) | 304 | 149 | 31 | 484
    Caucasian | 261 | 120 | 25 | 406
    Hispanic or Latino: number analyzed (Participants) | 304 | 149 | 31 | 484
    Hispanic or Latino | 15 | 8 | 0 | 23
    Native Hawaiian or other Pacific Islander: number analyzed (Participants) | 304 | 149 | 31 | 484
    Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
    Other: number analyzed (Participants) | 304 | 149 | 31 | 484
    Other | 0 | 1 | 0 | 1
    Not disclosed: number analyzed (Participants) | 304 | 149 | 31 | 484
    Not disclosed | 6 | 7 | 0 | 13
Region of Enrollment [Count of Participants; unit: Participants] — Data is based on all available data. Population: More subjects in the "Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study" Arm/Group completed the Baseline outcome measure and Region of Enrollment (359) than the Age and Sex Baseline measures which had 298 patients and the Race/Ethnicity which had 304.
  Participants
    United States | 359 | 149 | 31 | 539
Overall Pain Numeric Rating Scale (NRS) at Baseline [Mean (Standard Deviation); unit: units on a scale] — The Numeric Rating Scale is a tool for patient self-reporting of pain. The scale consists of 11 points, ranging from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable" Population: Data is based on all available data.
  units on a scale
    number analyzed (Participants) | 359 | 148 | 30 | 537
    (all) | 5.9 (2.3) | 7.6 (1.6) | 7.3 (1.4) | 6.5 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Pain Responder Rate
Description: Proportion of subjects with 50% or greater reduction in Low Back pain
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Boston Scientific SCS Systems (Day 0 Enrollment): All commercially approved Boston Scientific neurostimulation systems indicated for the treatment of chronic pain, except for Precision™ and Precision™ Plus.
  Neurostimulation System: Spinal cord stimulation
- Boston Scientific SCS Systems (Day 0 SCS Trial Procedure); Boston Scientific SCS Systems (Day 0 IPG Activation): All commercially approved Boston Scientific neurostimulation systems indicated for the treatment of chronic pain.
  Neurostimulation System: Spinal cord stimulation
Arm/Group | Boston Scientific SCS Systems (Day 0 Enrollment) | Boston Scientific SCS Systems (Day 0 SCS Trial Procedure) | Boston Scientific SCS Systems (Day 0 IPG Activation)
Number analyzed (Participants) | 215 | 67 | 29
Participants | 158 | 49 | 21

ADVERSE EVENTS:
Time Frame: From the time a subject sign the study Informed Consent through 3-year visit (NAVITAS), 4-year visit (ENVISION) or study withdrawal.
Description: Other (Not including Serious) Adverse Events definition differs from clinicaltrials.gov results Data Element definition - Per the study protocol, only device hardware and/or procedure related adverse events were monitored/assessed. Other, non-serious adverse events not related to the device hardware and/or procedure were not collected or assessed in this study.
  All Serious Adverse Events and All-Cause Mortality were monitored/assessed per the clinicaltrials.gov definition.
Arm/Group | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 SCS Trial Procedure) Navitas Study | Boston Scientific SCS Systems (Day 0 Implantable Pulse Generator (IPG) Activation) Navitas Study
All-Cause Mortality (participants affected / at risk) | 3/363 | 0/150 | 0/31
Serious Adverse Events (participants affected / at risk) | 51/363 | 16/150 | 12/31
Other Adverse Events (participants affected / at risk) | 0/363 | 0/150 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study (N=363) | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 SCS Trial Procedure) Navitas Study (N=150) | Boston Scientific SCS Systems (Day 0 Implantable Pulse Generator (IPG) Activation) Navitas Study (N=31)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Pneumonia (Infections and infestations) | 4 (5) | 1 (1) | 2 (2) — Not related to device and procedure
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) — Not related to device and procedure
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Not related to SCS device and procedure
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) — Not related to device and procedure
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Not related to device and procedure
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) — Not related to device and procedure
Spinal decompression (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Not related to device and procedure
Implant site infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Not related to device and procedure
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Not related to device and procedure
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Not related to device and procedure
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Not related to device and procedure
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) — Not related to device and procedure
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Not related to device and procedure
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Not related to device and procedure
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) — Not related to device and procedure
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Not related to device and procedure
Postoperative wound infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) — Not related to device and procedure
Empyema (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) — Not related to device and procedure
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Incision site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Not related to device and procedure
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Not related to device and procedure
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Pulmonary oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Hypertensive heart disease (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) — Not related to device and procedure
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Peripheral nerve lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Spinal epidural haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Wrist fracture (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Malnutrition (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) — Not related to device and procedure
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Medical device pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to device and procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 Enrollment) ENVISION Study (N=363) | Boston Scientific Spinal Cord Stimulator (SCS) Systems (Day 0 SCS Trial Procedure) Navitas Study (N=150) | Boston Scientific SCS Systems (Day 0 Implantable Pulse Generator (IPG) Activation) Navitas Study (N=31)
Implant site pain (General disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT03240588/Prot_SAP_000.pdf